CLINICAL TRIAL: NCT01182272
Title: Proof-of-Concept Phase II Study to Evaluate the Anti-Tumor Activity of Sorafenib Along With Pathological and Molecular Changes in Tumor Samples From Patients With Resectable Hepatocellular Carcinoma
Brief Title: Sorafenib Tosylate in Treating Patients With Liver Cancer That Can Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000682840; FRE-GERCOR-D09-1-BIOSHARE; EUDRACT-2009-018058-44; EU-21058
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized resectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Sorafenib; Neoadjuvant Therapy

INTERVENTIONS:
Drug: sorafenib tosylate
Other: laboratory biomarker analysis
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sorafenib tosylate works in treating patients with liver cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess anti-tumor activity of neoadjuvant sorafenib tosylate in tumor samples from patients with resectable hepatocellular carcinoma (HCC).

Secondary

* To characterize pathologic findings in sorafenib tosylate pre-treated patients undergoing surgical resection for HCC: 1-2 core tumor biopsies will be performed prior to treatment and at day 35.
* To evaluate the number of R0 resections in these patients.
* To correlate pathological biomarker changes in resected tumors after 4-week treatment with sorafenib tosylate in comparison with biopsies obtained prior to treatment in these patients.
* To evaluate plasma biomarkers, including PIGF, VEGF-A, VEGF-C, sVEGFR2, sVEGFR3, sKIT, IL-6, Ang2, IL-8, bFGF, AFP, collagen 4, endostatin, thrombospondin, TSP-1 and angiostatin, and CXCL12 at baseline, day 28, and the day before surgery.
* To identify potential biomarkers of sensitivity and/or resistance on biological and pathological samples of these patients (exploratory).
* To characterize the safety profile of sorafenib tosylate in these patients.
* To assess the tolerance of liver resection after sorafenib tosylate treatment of these patients.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib tosylate twice daily on days 1-28 in the absence of unacceptable toxicity. Approximately 7 days after completion of sorafenib tosylate therapy, patients undergo liver resection.

Blood and tissue specimens are collected periodically for laboratory and biomarker assessments. Biomarkers include both molecular markers investigating the direct antitumor effects of sorafenib tosylate against cancer cells vs the effects of the drug on angiogenesis.

After completion of study treatment, patients are followed up on day 50 and at 3 months after surgery.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatocellular carcinoma (HCC)

  * Fibrolamellar or mixed histology allowed
  * No cholangiocarcinoma or other tubal disease
* Must be eligible for conservative hepatic resection or liver resection with curative intent
* No cirrhosis with Child-Pugh score > 7
* Chronic liver disease without liver insufficiency and without portal liver hypertension allowed
* No known history or presence of metastatic brain or meningeal tumors

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* WBC > 3,000/µL
* ANC > 1,500/µL
* Platelet count ≥ 100,000/µL
* Hemoglobin ≥ 9 g/dL
* Bilirubin < 1.5 times upper normal limit (ULN)
* AST and ALT ≤ 5 times UNL
* Alkaline phosphatase ≤ 5 times ULN
* Serum creatinine < 2 times ULN
* PT/INR/PTT < 1.5 times UNL
* Amylase and lipase < 1.5 times ULN
* Negative pregnancy test
* Fertile patients must use effective contraception
* Body mass index 18.5-30 kg/m^2 (WHO normal range: 18.5-25 kg/m^2)
* Able to swallow oral compound
* No criterion for unresectability or medical condition that contraindicates surgical resection
* No serious concurrent systemic disorder incompatible with the study, including any of the following:

  * Uncontrolled hypertension (i.e., BP > 150/100 mm Hg despite optimal therapy)
  * Active uncontrolled infection
  * Active alcoholism
* No prior medical disorder, including any of the following:

  * Cardiac arrhythmias requiring anti-arrhythmics (excluding beta-blockers or digoxin for chronic atrial fibrillation)
  * Active coronary artery disease or ischemia
  * Myocardial infarction within the past 6 months
  * NYHA class III-IV congestive heart failure
  * Pulmonary embolism within the past 6 months
  * Gastrointestinal bleeding within the past 6 months
* No other prior malignancy within the past 5 years, except basal cell or squamous cell skin carcinoma or cured in situ cervical carcinoma
* No history or concurrent seizure disorder requiring medications (e.g., antiepileptic drugs)
* No history of HIV infection, or chronic hepatitis B or C
* No active clinically serious bacterial or fungal infection (i.e., grade 2 CTCAE v. 3)
* No condition that is unstable or could jeopardize the safety of the patient and his/her compliance with the study
* No substance abuse or medical, psychological, or social condition that could interfere with adherence to the study
* No known or suspected allergy to the investigational agent or to any agent given concurrently
* No presence of asthenia or rash > CTC grade 1 at enrollment
* Must be registered in a national health-care system

PRIOR CONCURRENT THERAPY:

* No prior orthotopic liver transplantation
* Not a candidate for orthotopic liver transplantation
* No prior systemic or loco-regional treatment for HCC
* No prior organ allograft
* No treatment with any other investigational medicinal product within the past 28 days
* No concurrent treatment with full-dose anticoagulants

  * Deep-vein or catheter-associated thrombosis prophylaxis allowed
  * Warfarin or heparin therapy allowed if the coagulation parameters were within the acceptable ranges prior to initiation of anticoagulant therapy
* No concurrent or chronic co-administration of CYP3A4 inducers (e.g., rifampin, Hypericum perforatum, phenytoin, carbamazepine, phenobarbital, or dexamethasone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Antiangiogenic effects of sorafenib tosylate
Significant pathological changes

SECONDARY OUTCOMES:
Pathologic findings in sorafenib tosylate pre-treated patients undergoing surgical resection for hepatocellular carcinoma
Number of R0 resections
Correlations between baseline patient characteristics, cancer biomarkers, and outcome variables and resected tumors
Plasma biomarkers at baseline, day 28, and the day before surgery
Safety profile of sorafenib tosylate
Tolerance of liver resection after sorafenib tosylate treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Faivre, Principal Investigator — Hopital Beaujon
Locations (1):
- Hopital Beaujon, Clichy, France